CLINICAL TRIAL: NCT05208190
Title: Clozapine for the Prevention of Violence in Schizophrenia: a Randomized Clinical Trial
Acronym: REVISIT-C
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ragy Girgis, Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I20-02054; 1R01MH120317-01A1 (NIH)
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Clozapine; Therapeutics

STUDY DESIGN:
Intervention Model Description: single-blind, open-label, randomized, active comparator (TAU) controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Blinded raters and a blinded adjudication committee to ensure that the outcome is valid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Clozapine (Experimental): treatment with clozapine naturalistically administered (as per clinical guideline).
  Interventions: Drug: Clozapine
- Treatment as usual (Active Comparator): open label naturalistic treatment as usual with any antipsychotic other than clozapine
  Interventions: Drug: treatment as usual

INTERVENTIONS:
Drug: Clozapine — treatment will occur naturalistically, as per standard clinical guidelines
  Other Names: clozaril
  Arms: Clozapine
Drug: treatment as usual — naturalistic treatment with any other antipsychotic medication except clozapine
  Arms: Treatment as usual

SUMMARY:
Two-hundred and eighty individuals with schizophrenia who have a recent history of violent acts will be randomized in this 2-arm, parallel-group, 24-week, open-label, 7-site clinical trial to examine the effects of treatment with clozapine vs antipsychotic treatment as usual (TAU) for reducing the risk of violent acts in real-world settings

DETAILED DESCRIPTION:
This is a single-blind, open-label, randomized, active comparator (TAU) controlled clinical trial to examine the effects of clozapine vs. TAU on the risk for violent acts as measured by the MacArthur Community Violence Interview (MCVI) and to examine the effects of clozapine vs. TAU on the Excitement Factor of the PANSS. Adults age 18-65 with schizophrenia or schizoaffective disorder who have committed a violent act within 6 months and are appropriate for treatment with clozapine or TAU will receive treatment for 24 weeks which will be naturalistically administered. Participants will also participate in assessments and appropriate medical monitoring which will include blood draws, pharmacokinetic blood samples, and physical exams, etc. Cox proportional hazards survival modeling will be used to test the association between treatment group and time until first violent act after randomization (i.e., number of weeks form randomization to violent act).

The NYSPI site is currently paused and has been paused since an institutional pause on human subjects research began in June, 2023. (The IO in concurrence with the IRB paused human subjects research on June 12, 2023. The U.S. Department of Health and Human Services (HHS) Office of Human Research Protections (OHRP) issued an FWA restriction on NYSPI research that also included a pause of human subjects research as of June 23, 2023.) Therefore, the NYSPI site is not enrolling at this time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual-5 (DSM-5) diagnosis of schizophrenia or schizoaffective disorder by the Structured Clinical Interview for DSM-5 (SCID-5)
* commission of a minor or serious act of violence as measured by the MCVI in the last six months
* willing and able to provide informed consent
* medically stable in judgment of physician providing study treatment
* appropriate for treatment with either clozapine or TAU, i.e., that there is clinical equipoise between the two treatment options. Individuals who are currently medication free or on any antipsychotic, with the exception of clozapine or long-acting injectable medication with a dosing interval of more than 30 days will be eligible

Exclusion Criteria:

* An unstable of serious medical or neurological condition including a myeloproliferative disorder or condition that surprises the bone marrow
* A history of intolerance/allergy to clozapine (e.g., agranulocytosis, small bowel obstruction, or myocarditis)
* A history of intellectual impairment
* pregnant or lactating women; women who are able to become pregnant but who are not willing to sue effective methods of birth control
* Individuals who score a 3, 4, or 5 within the previous month on the suicidal ideation section of the Columbia Suicide Severity Rating Scale (CSSRS), have any suicidal behavior (not including Not Suicidal Self Injury) within the previous 3 months, or are, in the opinion of the investigator, at too high of a risk for suicide to be safety treated in a randomized trial in which they may not be treated with clozapine
* Documented intolerance to or lack of any therapeutic benefit with clozapine after a full trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness outcome: Violent acts | Time to violent act from randomization to treatment completion (24 weeks)
  violent acts as measured by the MacArthur Community Violence Interview
Target engagement outcome: Excitement Factor of the Positive and Negative Syndrome Scale (PANSS) | Randomization to end of study treatment (24 weeks)
  a composite of the scores of excitement, uncooperativeness, poor impulse control, and hostility)

SECONDARY OUTCOMES:
Effect on aggression | Randomization to end of treatment (24 weeks)
  examine the effects of clozapine vs TAU on aggression as measured by the Point Subtraction Aggression Paradigm
Positive symptoms and substance use | Randomization to end of treatment (24 weeks)
  explore effects of clozapine vs TAU on the positive symptom sub scale of the PANSS and alcohol and illicit substance use, how these effects influence the risk for violent acts, and the degree to which clozapine's effects on the Excitement Factor of the PANSS are independent of its effects on total positive symptoms and substance use.

OTHER OUTCOMES:
Interventions to Prevent Violence | Randomization to end of treatment (24 weeks)
  examine the effects of clozapine vs TAU on interventions to prevent violence based on a querying clinicians treating patients about interventions to prevent violence at weeks 4, 8, 16 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Ragy Girgis, MD, Principal Investigator — New York State Psychiatric Institute
Locations (7):
- United States (7):
  - University of California, Los Angeles, Los Angeles, California
  - Augusta University Research Institute, Inc., Augusta, Georgia
  - University of Maryland School of Medicine, Baltimore, Maryland
  - NYU Langone Medical Center, New York, New York
  - New York State Psychiatric Institute, New York, New York
  - Manhattan Psychiatric Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina